CLINICAL TRIAL: NCT03137160
Title: An Open-Label, Proof-of-Concept Study of Ixekizumab in the Treatment of Pyoderma Gangrenosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Ben H Kaffenberger, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017H0045
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ixekizumab (Taltz) (Experimental): We have received funding for only a small pilot study to prove a benefit from Interleukin-17 inhibition in Pyoderma Gangrenosum . Therefore, there is only one treatment arm. The primary outcome will be a comparison of week 12 to baseline regarding a two-point improvement in the Investigator Global Assessment.
  Interventions: Biological: Ixekizumab

INTERVENTIONS:
Biological: Ixekizumab — Injection
  Other Names: Taltz

SUMMARY:
An Open-Label, Proof-Of-Concept, Study of Ixekizumab in the Treatment of Pyoderma Gangrenosum

DETAILED DESCRIPTION:
This is a Phase II study that will be open label and include a total of five patients who will receive the investigational product. These patients will have histological testing to rule out competing etiologies and require 3rd party adjudication/confirmation on agreement of the diagnosis. These patients will undergo 12 weeks of ixekizumab dosed every 2 weeks with follow-up until week 16.

ELIGIBILITY:
Inclusion Criteria:

* Major inclusion criteria:
* Have a clinical diagnosis of classic Pyoderma Gangrenosum for at least 3 months as determined by the investigator and an external reviewer on the basis of results from clinical, histological and laboratory assessments
* At screening, have a Pyoderma Gangrenosum ulcer characterized by 'item a' AND 3/5 features in 'item b' OR 2/5 features in 'item b' with support from one of the conditions listed in c.

  a. Stable or increasing size within 2 months preceding screening by patient report or documentation b. Features such as violaceous border, undermining, d. Intralesional corticosteroids within 8 weeks of day 0; topical immunomodulators are permitted.

  e. Wound debridement within 2 weeks of Day 0; dressing changes allowed per investigator discretion.

  g. Systemic antibiotics within 2 weeks of Day 0 h. Live, attenuated vaccines within 3 months of Day 0; or live, seasonal-flu- or H1N1 vaccines within 2 weeks of Day 0. Note: recombinant- and/or killed vaccines are permitted.

  i. Hyperbaric treatment within 4 weeks of Day 0 j. Investigational drug or investigational device within 30 days or 5 half-lives of Day 0, whichever is longer k. Prior exposure to ixekizumab l. Other treatments not described above should be maintained at a stable dose and frequency throughout the study as best as possible 13. Major, general surgery within 3 months of screening, or anticipated general surgery during the study period 14. Pregnancy, plans to become pregnant during the course of the study, delivery within 3 months of screening, or breast-feeding 15. If previous use of cyclosporine or systemic corticosteroids, failure to have any stabilization/response is exclusionary. This potentially indicates the disease is not Pyoderma Gangrenosum.

Exclusion Criteria:

* Major exclusion criteria:

  1. Any condition (e.g., psychiatric illness, severe alcoholism, or drug abuse) or situation that may compromise the ability of the subject to give written informed consent, may put the subject at significant risk, may jeopardize the subject's safety after exposure to the study drug, may confound the study results, or may interfere significantly with the subject's participation in the study
  2. History of malignancy within 2 years of screening other than carcinoma in situ of the cervix or adequately treated, non-metastatic, squamous or basal cell carcinoma of the skin
  3. History of seropositivity for HIV antibody; active or carrier status of hepatitis B [surface antigen (HBsAg) positive, or core antibody (anti-HBc) positive with negative surface antibody]; active hepatitis C (i.e. not treated or not cleared spontaneously, as confirmed by HCV PCR)
  4. History of severe allergic or anaphylactic reaction to monoclonal antibodies
  5. Systemic infection (excluding wound colonization) requiring oral antibiotics within 2 weeks of Day 0
  6. History of the following treatments:

     1. Anti-Tumor Necrosis Factor or other biologic therapies within 5 half-lives of screening
     2. Changes (addition, discontinuation, or changes in dose) in immunosuppressive medication (including cyclosporine, azathioprine, methotrexate, mycophenolate mofetil, apremilast, dapsone, or corticosteroids) within 2 months of Day 0
     3. Systemic corticosteroids > 20 mg per day (prednisone or prednisone equivalent) within 8 weeks of Day 0, or change in dose within 8 weeks of Day 0. Steroids may be tapered (although not increased above the Day 0 dose) during the trial as determined by the investigator.

they are prescribed at stable doses for two months prior to baseline and are 20 mg or less per day of prednisone or other equivalently-dosed corticosteroids.

4. Intralesional corticosteroids within 4 weeks of screening and during the study are not permitted 5. Other therapies that are non-immunosuppressive and non-investigational can be started or continued at physician discretion provided the medicine has no history of association with progressive multifocal leukoencephalopathy. Antibiotics may be used as needed for evidence of superinfection, positive culture results, malodor, green discharge, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kaffenberger, MD, Principal Investigator — Dermatologist
Locations (1):
- The Ohio State University Dermatology, Gahanna, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study will be conducted in Columbus, OH, at The Ohio State University (OSU) dermatology clinical trials center. Both the principal investigator and the OSU dermatology center have extensive experience with industry-sponsored clinical trials in PG, having completing two trials in 2015-16
Pre-assignment Details: These patients will have histological testing to rule out competing etiologies and require 3rd party adjudication/confirmation on agreement of the diagnosis
Period: Overall Study
Arm/Group | Ixekizumab (Taltz)
Started (One screen failed due to infection and never enrolled or received drug) | 4
Completed | 2
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: These are patients who have been seen by the primary investigator with the diagnosis of pyoderma gangrenosum, typically within Ohio, USA
Arm/Group | Ixekizumab (Taltz)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants] — Age collected from medical records and confirmed with patient
  Participants
    <=18 years | 0
    Between 18 and 65 years | 4
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 49.5 [23 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number meeting criteria for inclusion [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Achieving 2-point Reduction in the 5-point Investigator Global Assessment (IGA) for the Target Ulcer at Week 12
Description: The primary outcome will be the proportion of subjects achieving a 2-point reduction in the 5-point investigator global assessment for the target ulcer at Week 12. The measure type and unit of measure are the proportion of participants.
  The IGA utilizes a 5 point Investigator Global Assessment measuring disease severity from 0- clear, 1-minimal, 2-mild, 3-moderate, 4- severe. 4 is the worst
Time Frame: 12 Weeks
Population: The proportion of subjects achieving a two point reduction in the five-point investigator global assessment (IGA) for the target ulcer from baseline to week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab (Taltz)
Number analyzed (Participants) | 4
Participants | 0
Statistical Analysis 1: Comparison: Ixekizumab (Taltz); This is the Investigator Global Assessment comparing the proportion of subjects who achieved a 2 pt reduction at study close (0); Test type: Superiority; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 16 weeks per patient and 1 year for the trial. Patient 01: data collected for 16 weeks. Patient EOT at week 16 Patient 02: Data collected for 2 weeks. Lost to FU after week 2 Patient 03: data collected for 6 weeks. Patient EOT visit at week 6 Patient 04: data collected for 6 weeks. EOT visit at week 6
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Ixekizumab (Taltz)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab (Taltz) (N=4)
sepsis (Blood and lymphatic system disorders) | 1 (1) — Sepsis due to LLE wound infection
infection (Infections and infestations) | 1 (1) — Bilateral Infection of Pyoderma Gangrenosum
sepsis (Blood and lymphatic system disorders) | 1 (1) — Severe Sepsis secondary to Pneumonia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab (Taltz) (N=4)
hypotension (Cardiac disorders) | 2 (2)
fever (Immune system disorders) | 2 (3)
vomitting (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (2)
infection of ulcer (Infections and infestations) | 1 (1)
pneumonia (Immune system disorders) | 1 (1)
h influenza (Immune system disorders) | 1 (1)
low WBC (Infections and infestations) | 1 (1)
low igG levels (Immune system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial stopped early due to safety. Patients were all previously hospitalized as well. High risk of re-hospitalization was not necessarily unexpected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT03137160/Prot_SAP_001.pdf